CLINICAL TRIAL: NCT03110042
Title: High Versus Low SpO2 Oxygen Therapy in Patients With Acute Heart Failure
Brief Title: HILO-HF Registry: High Versus Low SpO2 Oxygen Therapy in Patients With Acute Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: HILO-HF Registry
Record Dates: First submitted 2017-04-01; First posted 2017-04-12 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: All patients will receive usual standard of care with the heart failure management including the routine supplemental oxygen therapy.

SUMMARY:
The HILO-HF Registry is a single centre registry that will be performed to provide information on the usual baseline oxygen saturation (SpO2) in patients presenting to ED with a primary ED diagnosis of AHF

ELIGIBILITY:
Inclusion Criteria:

* Patients >40 years of age presenting to the ED with AHF
* With or without tested BNP
* With or without admission to hospital for treatment of HF\
* Patients must be recruited within the first 24 hours of presenting to the ED.

Exclusion Criteria:

* Patients on home oxygen
* Patients with known prior hypercapnic failure (PaCO2>50 mmHg)
* Asthma
* Primary pulmonary hypertension
* Patients requiring urgent positive pressure ventilation or intubation or on >10 L/min oxygen

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >40 years of age presenting to the ED with AHF
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in blood oxygen saturation levels from baseline to 72 hours | 72 hours

SECONDARY OUTCOMES:
Dyspnea on visual analogue scale (VAS) to 72 hours | 72 hours
Change in global symptoms using Patient Global Assessment (PGA) measure to 72 hours | 72 hours
Change in Peak Expiratory Flow | 72 hours
Rate of patients with Worsening Heart Failure | 7 days
30-day composite clinical event (all-cause mortality, HF readmission, days alive and out of hospital) | 30days

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital / Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada